CLINICAL TRIAL: NCT04548700
Title: Clinical Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of Liposomal Mitoxantrone Hydrochloride Injection Combined With Cyclophosphamide, Vincristine and Prednisone in the Treatment of Untreated PTCL
Brief Title: Liposomal Mitoxantrone Hydrochloride Injection,Cyclophosphamide, Vincristine and Prednisone in the Treatment of PTCL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor has adjusted its R&D strategy.
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-011
Record Dates: First submitted 2020-08-28; First posted 2020-09-14 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2020-08

CONDITIONS: Treatment-naïve; Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Cyclophosphamide; Vincristine; Prednisone; PART-1 RNA, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-finding and dose-expansion (Experimental): Dose-finding stage: Patients with treatment-naïve PTCL will receive sequentially higher doses of liposomal mitoxantrone hydrochloride in combination with Cyclophosphamide, Vincristine and Prednisone for 6 cycles (planned) (28 days per cycle). The initial dose of liposomal mitoxantrone hydrochloride is 12 mg/m2.
  Dose-expansion stage: Patients with treatment-naïve PTCL will receive liposomal mitoxantrone hydrochloride at RP2D in combination with Cyclophosphamide, Vincristine and Prednisone for 6 cycles (planned) (28 or 21 days per cycle).
  Interventions: Drug: Dose-finding stage: Liposomal mitoxantrone hydrochloride, Cyclophosphamide, Vincristine and Prednisone; Drug: Dose-expansion stage: Liposomal mitoxantrone hydrochloride, Cyclophosphamide, Vincristine and Prednisone

INTERVENTIONS:
Drug: Dose-finding stage: Liposomal mitoxantrone hydrochloride, Cyclophosphamide, Vincristine and Prednisone — Drug: Liposomal mitoxantrone hydrochloride (12 mg/m2, 15 mg/m2, 18 mg/m2) will be administered by an intravenous infusion on day 1 of each 28-day cycle.
  Drug: Cyclophosphamide (750 mg/m2) will be administered by an intravenous infusion on day 1 of each 28-day cycle.
  Drug: Vincristine (1.4 mg/m2 with 2 mg as the maximum dose) will be administered by an intravenous injection on day 1 of each 28-day cycle.
  Drug: Prednisone (100 mg/d) will be taken orally from day 1 to day 5 of each 28-day cycle.
  Other Names: Part1
Drug: Dose-expansion stage: Liposomal mitoxantrone hydrochloride, Cyclophosphamide, Vincristine and Prednisone — Drug: Liposomal mitoxantrone hydrochloride (at RP2D) will be administered by an intravenous infusion on day 1 of each 28- or 21-day cycle.
  Drug: Cyclophosphamide (750 mg/m2) will be administered by an intravenous infusion on day 1 of each 28- or 21-day cycle.
  Drug: Vincristine (1.4 mg/m2 with 2 mg as the maximum dose) will be administered by an intravenous injection on day 1 of each 28- or 21-day cycle.
  Drug: Prednisone (100 mg/d) will be taken orally from day 1 to day 5 of each 28- or 21-day.
  Other Names: Part2

SUMMARY:
This is a multicentre, open-label, single-arm, phase Ib clinical study to evaluate the safety, tolerability, efficacy and pharmacokinetics of liposomal mitoxantrone hydrochloride in combination with Cyclophosphamide, Vincristine and Prednisone in the frontline treatment of patients with peripheral T cell lymphoma (PTCL).

DETAILED DESCRIPTION:
The study is to investigate the safety, tolerability, efficacy and pharmacokinetics of liposomal mitoxantrone hydrochloride in combination with Cyclophosphamide, Vincristine and Prednisone in the frontline treatment of patients with PTCL by conducting in two stages, Dose-finding stage and Dose-expansion stage.In Dose-finding stage, patients with treatment-naïve PTCL will be assigned to receive sequentially higher doses of liposomal mitoxantrone hydrochloride ranging from 12 to 18 mg/m2 plus Cyclophosphamide, Vincristine and Prednisone (28 days per cycle). The dose escalation will follow the classic 3+3 design. The recommended Phase 2 dose (RP2D) of liposomal mitoxantrone hydrochloride will be determined according to the Dose-finding results. In Dose-expansion stage, additional patients will be recruited into two groups, the Q4W group（28 days per cycle）and the Q3W group（21 days per cycle）, to receive liposomal mitoxantrone hydrochloride at the RP2D combined with Cyclophosphamide, Vincristine and Prednisone. All patients will receive the treatment for the planned 6 cycles or until disease progression or unacceptable drug-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent
2. Age ≥18, ≤70years, no gender limitation
3. Histologically confirmed diagnosis of treatment-naïve PTCL. Eligible histologies are limited to the following: Peripheral T-cell lymphoma - not otherwise specified (PTCL-NOS),Angioimmunoblastic T-cell lymphoma (AITL), ALK -positive Anaplastic Large cell Lymphoma（ALCL）, ALK-negative ALCL; Other PTCL that investigators consider to be appropriate to be enrolled
4. PTCL with fluorodeoxyglucose (FDG) avidity that can be evaluated by PET/CT
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1
6. The following required baseline laboratory data: Absolute neutrophil count (ANC) ≥1.5×109/L, Platelet count (PLT) ≥75×109/L, Hemoglobin(HB)≥ 80g/L, Total bilirubin (TBIL) ≤1.5X upper limit of normal (ULN) , Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5X ULN , Serum creatinine (Scr) ≤1.5X ULN
7. Females of childbearing potential must have a negative serum beta human chorionic gonadotrophin (β-hCG) pregnancy test result prior to enrollment and must agree to use an effective contraception method for the duration of the study treatment and 12 months after the last dose of study therapy
8. Males of reproductive potential must agree to use an effective contraceptive method for the duration of the study treatment and 12 months after the last dose of study therapy

Exclusion Criteria:

1. Current diagnosis of any of the following: extranodal natural killer/T-cell lymphoma, nasal type(NKTCL), Mycosis fungoides (MF)/ Sézary syndrome (SS), Primary cutaneous ALCL，and Adult T-cell leukemia/lymphoma
2. Leukemic phase of lymphoma (≥20% lymphoma cell in the bone marrow), or central nervous system (CNS) involvement, or hemophagocytic syndrome
3. Life expectancy < 6 months
4. History of allergy to anthracyclines or liposomes
5. History of contraindications to cyclophosphamide, vincristine or prednisone
6. Prior anti-lymphoma therapy except short-term or low-dose corticosteroid treatment
7. Impaired cardiac function or significant cardiac disease
8. Positive test results for HBsAg antigen and HBV-DNA, or hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) antibody
9. Major surgery within 4～6weeks prior to screening. Or have a surgical schedule during the study
10. A serious infection within 4 weeks prior to screening and not suitable for the study according to the judgment of the investigator
11. Uncontrolled hypertension at screening
12. Uncontrolled diabetes at screening
13. History of active visceral hemorrhage in the recent 3 months prior to screening
14. History of other tumors in the past five years prior to screening. Patients with curable tumors (such as skin basal cell carcinoma, carcinoma in situ of the cervix or of the breast, intramucosal carcinoma in situ of the gastrointestinal tract or localized prostate cancer) could be enrolled after completely cured
15. History of solid organ transplantation
16. Known psychiatric disorders or cognitive disorder
17. Known alcohol or drug abuse
18. Pregnant or breastfeeding women
19. Not suitable for this study as determined by the investigator due to other reasons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Dose-finding stage: The incidence of dose limited toxicities (DLTs) | Cycle 1 (28 days)
  To identify the DLTs
Dose-finding stage:The incidence of AE and SAE | up to 24 weeks
  To identify the incidence of AE and SAE, abnormalities in clinical laboratory assessments, ECGs, echocardiography, vital sign assessments, and physical exams
Dose-expansion stage: The incidence of AE and SAE | up to 18-24 weeks
  To identify the incidence of AE and SAE, abnormalities in clinical laboratory assessments, ECGs, echocardiography, vital sign assessments, and physical exams

SECONDARY OUTCOMES:
Dose-finding stage: complete response(CR) rate | up to 24 weeks
  To investigate the preliminary antitumor efficacy
Dose-finding stage: duration of complete response（DoCR） | Throughout study completion,an average of 18 months
  To investigate the preliminary antitumor efficacy
Dose-finding stage: overall response rate (ORR) | up to 24 weeks
  To investigate the preliminary antitumor efficacy
Dose-finding stage: progression-free survival（PFS） | Throughout study completion,an average of 18 months
  To investigate the preliminary antitumor efficacy
Dose-finding stage：the pharmacokinetic parameters Cmax | Cycle 1 to Cycle 6(each cycle is 28 days)
  To investigate the PK characteristics
Dose-finding stage：the pharmacokinetic parameters AUC0-t | Cycle 1 to Cycle 6(each cycle is 28 days)
  To investigate the PK characteristics
Dose-expansion stage: CR rate | up to 24 weeks
  To investigate the preliminary antitumor efficacy
Dose-expansion stage: DoCR | Throughout study completion,an average of 18 months
  To investigate the preliminary antitumor efficacy
Dose-expansion stage: ORR | up to 18-24 weeks
  To investigate the preliminary antitumor efficacy
Dose-expansion stage: PFS | Throughout study completion,an average of 18 months
  To investigate the preliminary antitumor efficacy
Dose-expansion stage: the pharmacokinetic parameters Cmax | Cycle 1(each cycle is 21or28 days)
  To investigate the PK characteristics
Dose-expansion stage: the pharmacokinetic parameters AUC0-t | Cycle 1(each cycle is 21or28 days)
  To investigate the PK characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiang Huang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China